CLINICAL TRIAL: NCT00064610
Title: A Phase I/II, Open Label, Dose Escalation Study to Determine the Tolerance and Preliminary Activity of PS-341 Plus Docetaxel in Patients With Advanced Androgen-Independent Prostate Cancer Requiring Chemotherapy
Brief Title: Phase I/II Dose Escalation Study of VELCADE® and Docetaxel in Patients With Advanced Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M34101-033
Record Dates: First submitted 2003-07-10; First posted 2003-07-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Prostatic Neoplasms
Keywords: Advanced androgen-independent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bortezomib; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: VELCADE TM (bortezomib) for Injection

SUMMARY:
The purpose of this study is to evaluate how safe PS-341(VELCADE) is when given with Docetaxel (Taxotere) to patients with androgen-independent prostate cancer, and also to see what effects (good and bad) it has on you and on your cancer.

DETAILED DESCRIPTION:
This is a dose escalation study, which means that the first group of patients will receive a low dose of PS-341 (VELCADE) and Docetaxel (Taxotere). If the low dose of VELCADE and Taxotere appears to be safe, then the next group of patients will receive a higher dose of VELCADE and Taxotere.

ELIGIBILITY:
Inclusion criteria

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Patient has histologically-confirmed advanced and/or metastatic androgen-independent prostate cancer requiring anti-neoplastic treatment.
* Previous or concurrent hormone therapy with a luteinizing hormone-releasing hormone analog (e.g., leuprolide) does not preclude enrollment in the study.
* Patient has progressive measurable or evaluable disease, defined as meeting at least one of the following three criteria [1]:

  1. Progressive measurable disease (changes in the size of lymph nodes or parenchymal masses on physical examination or x-ray).
  2. Progressive bone metastasis [presence of new lesion(s) on a bone scan].
  3. Progressive PSA, as evidenced by two separate measurements taken at least one week apart and confirmed by a third, and if necessary, a fourth measurement.

     * If the third measurement is not greater than the second measurement, then a fourth measurement must be taken; the fourth measurement must be greater than the second measurement for the patient to be eligible for enrollment in the study.
     * The confirmatory PSA measurement (i.e., the third or, if applicable, fourth PSA measurement) must be greater than or equal to 5 ng/mL.
* Patient is 18 years of age or older.
* Patient has a Karnofsky performance status of 60% or greater.
* Patient has a life expectancy of three months or longer.
* Patient has all of the following pretreatment laboratory data within 14 days before the first study drug dose:
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mm3.
* Platelets greater than or equal to100,000/mm3.
* Hemoglobin >8.0 g/dL.
* Serum creatinine less than or equal to 2.5 mg/dL.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
* Patient agrees to use an acceptable barrier method for contraception from Screening through 90 days after the last study drug dose. [It is recommended that female partners of male patients enrolled in this study also use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence).]

Exclusion criteria Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Patient has received chemotherapy within four weeks, nitrosoureas within six weeks, or antibody therapy within eight weeks of enrollment.
* Patient has received radiation therapy within four weeks of enrollment.
* Patient has not recovered from all toxic effects of previous chemotherapy or radiation or antibody therapy.
* Patient received treatment with flutamide within four weeks of enrollment or nilutamide or bicalutamide within six weeks of enrollment.
* Patient has had any major surgery within four weeks of enrollment.
* Patient has a history of allergic reactions to diuretics or anti-emetics suggested to be administered in conjunction with study drug
* Patient has a history of severe hypersensitivity reaction to docetaxel or other agents formulated with polysorbate 80.
* Patient had a myocardial infarction within six months of enrollment or has uncontrolled angina, severe uncontrolled ventricular arrhythmias, symptomatic congestive heart failure, unstable angina pectoris, or electrocardiographic evidence of acute ischemia
* Patient has uncontrolled brain metastases or central nervous system disease.
* Patient has Grade 2 or higher peripheral neuropathy
* Patient has any of the following pretreatment laboratory data within 14 days before the first study drug dose:

  * Total bilirubin > than the upper limit of normal (ULN).
  * Alanine transaminase (ALT) and/or aspartate transaminase (AST) >1.5 x the ULN concurrent with alkaline phosphatase >2.5 x the ULN.
  * Alkaline phosphatase >5 x the ULN, unless shown by fractionation to be bone-derived and AST, ALT, bilirubin, gamma glutamyl transferase (GGT), and 5'nucleotidase are <1.5 x the ULN and bilirubin is within normal range.
  * Serum testosterone 50 ng/mL or higher.
* Patient is HIV-infected.
* Patient is hepatitis B surface antigen positive or has previously documented hepatitis C infection.
* Patient has an uncontrolled intercurrent illness (e.g., active infection).
* Patient has another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2002-12; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Columbia-Presbyterian Hospital, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee